CLINICAL TRIAL: NCT03045042
Title: Search for Serum/Plasma Biomarkers in Pompe's Disease
Acronym: BIOPOMPE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: IIBSP-BIO-2017-02; GZ-2015-11342 (Other: Genzyme)
Record Dates: First submitted 2017-01-27; First posted 2017-02-07 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Late Onset Pompe Disease; Pompe Disease
Keywords: Pompe; microRNA; biomarker; muscle MRI; glycogenosis
MeSH Terms: conditions — Glycogen Storage Disease Type II; Glycogen Storage Disease | interventions — GAA protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated patients: Patients with late onset Pompe disease treated with the enzyme replacement therapy
  Interventions: Drug: Enzyme Replacement Agent
- Non treated patients: Patients with late onset Pompe disease non treated with the enzyme replacement therapy

INTERVENTIONS:
Drug: Enzyme Replacement Agent — Patients will be treated following the decision of their doctors. The investigators are going to analyze serum samples of these patients
  Other Names: Myozyme
  Groups: Treated patients

SUMMARY:
This study aims to analyze serum and plasma samples from patients with late onset Pompe disease treated and not treated with enzyme replacement therapy (ERT) to identify microRNA that could be specific of the disease. The investigators will correlate the concentration of these microRNA with several muscle function tests and quantitative muscle MRI to know whether they are good biomarkers of progression.

ELIGIBILITY:
Inclusion Criteria:

* Genetic confirmation of Pompe disease

Exclusion Criteria:

* Pregnancy

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Late onset Pompe patiens
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
MicroRNA in serum samples | Baseline
  Investigators are going to study microRNA following a microarray analysis of serum samples from patients treated and non treated

SECONDARY OUTCOMES:
Muscle function test | Baseline and one year
  6 minutes walking test (6MWT), time to climb 4 steps, time to descend 4 steps, Activlim, time to walk 10 meter, Medical Research Council scale (MRC), myometry
Whole body muscle MRI | Baseline a and one year
  2 point dixon studies of thigh muscles
Changes in microRNA concentration | One year period
  Investigators will analyze concentration of microRNA after one year follow up in every single patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No